CLINICAL TRIAL: NCT02558647
Title: Overcoming Insomnia: A Large-scale Randomized Controlled Trial of Online Cognitive Behavior Therapy for Insomnia Compared With Online Patient Education About Sleep.
Brief Title: Overcoming Insomnia: Impact on Sleep, Health and Work of Online CBT-I
Acronym: NORSE-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Borge Sivertsen, Senior researcher, Norwegian Institute of Public Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFR:239985; HUNT-SHUTi (Other: Norwegian IPH; NTNU)
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Insomnia
Keywords: therapy; CBT-I; internet-based; online; short-term benefits; medium-term outcomes; health resource use; sick leave
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This is a parallel-group superiority RCT comparing internet-delivered CBT-I (a Norwegian language version of SHUTi) with online patient education about sleep (PE).
Who Masked: Participant, Investigator
Masking Description: Study participants are randomized to CBT-I or a potential active comparator (PE). Follow-up data is primarily self-report; data on sick leave etc is objective data obtained form national registers, with investigators are blinded to participant identity.
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT for insomnia (CBT-I) (Experimental): Internet-based cognitive-behavioral therapy for insomnia (CBT-I) comprises a fully automated, interactive, and tailored web-based program that incorporates the primary tenets of face-to-face CBT-I, including sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, and relapse prevention
  Interventions: Behavioral: CBT for insomnia (CBT-I)
- Psychoeducation about Sleep (PE) (Active Comparator): The PE intervention gives participants access to a website with information about insomnia symptoms; the impact, prevalence, and causes of insomnia; when to seek input from a doctor; and basic lifestyle, environmental, and behavioral strategies that may help to improve sleep.
  Interventions: Behavioral: Psycho-Education about Sleep (PE)

INTERVENTIONS:
Behavioral: CBT for insomnia (CBT-I) — CBT-I is an online, fully automated, interactive, and tailored web-based program that incorporates the primary tenets of face-to-face CBT-I, including sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, and relapse prevention.
  Other Names: SHUTi
  Arms: CBT for insomnia (CBT-I)
Behavioral: Psycho-Education about Sleep (PE) — PE provides online information about insomnia symptoms; the impact, prevalence, and causes of insomnia; when to seek input from a doctor; and basic lifestyle, environmental, and behavioral strategies that may help to improve sleep.
  Other Names: passive education/ sleep hygeine
  Arms: Psychoeducation about Sleep (PE)

SUMMARY:
Insomnia is a major public health concern. While cognitive behavior therapy for insomnia (CBT-I) is acknowledged as the best available intervention, there are unanswered questions about its wider dissemination, socio-economic benefits and its impact on health resource utilization. The aim of this randomized controlled trial (RCT) is to investigate the effectiveness of a fully automated online version of CBT-I compared with online patient education about sleep (PE). Outcome measures comprise changes in symptoms of insomnia, time off work due to sick leave, as well as medication and health resource utilization. Also, we will examine putative mediators and selected potential psycho-bio-social moderators of the effects of the intervention.

DETAILED DESCRIPTION:
This is a two-arm RCT that assesses the benefits of online CBT-I compared with an alternative, active control intervention (online patient education about sleep (PE)). We will randomize 1500 individuals and collect follow-up data for up to two years. First, we will examine any differential change in the severity of insomnia, immediately after completing the interventions. Secondly, we will examine if there are differential changes in symptoms of physical and mental health (e.g. psychological distress, fatigue, and health related quality of life) immediately post-intervention, and whether any improvements in insomnia or other symptoms are reported at further follow-ups (6- and 24 months post treatment termination). Third, we will use national registry data collected routinely in Norway to compare rates of time off work due to sick leave days for up to two years before and after participating in the RCT, as well as monitoring medication and health resource utilization according to condition in the same time interval. Fourth, we will try to extend the knowledge base about online interventions by undertaking exploratory analyses to assess whether change in specific clinical variables (e.g. sleep variability, psychological measures of beliefs about sleep) mediate the effects of the CBT-I intervention. Lastly, (subject to additional funding to collect saliva samples), we will examine a subset of psycho-bio-social factors to try to identify potential treatment moderators that might inform the stratification of individuals with insomnia into 'treatment-relevant' subgroups in the future (e.g. this may include also an exploration of 'therapygenetics').

ELIGIBILITY:
Inclusion criteria:

* Individuals aged >=18 years who score >= 12 on the Insomnia Severity Index (a score indicative of insomnia symptoms that significantly impact on individuals)
* Willing and able to give online informed consent.

Exclusion criteria:

* Individuals scoring >10 on the Epworth Sleepiness Scale (ESS) (which is suggestive of excessive daytime sleepiness) and/or answering that they usually or every day snore and stop breathing and have difficulties staying awake during the day (i.e., they positively endorse pre-selected indicators of sleep apnoea);
* Self-report of the presence of any medical conditions where a fully automated CBT-I may be contra-indicated (e.g. epilepsy, bipolar disorder, schizophrenia or psychotic disorders, and recent heart surgery)
* Participating in shift work.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index, ISI | Pre to 9 weeks post randomization (post treatment assessment)
  The ISI will be used to assess self-reported levels of insomnia severity. Range is 0-28. Higher values represent higher levels of insomnia symptom severity.

SECONDARY OUTCOMES:
Insomnia Severity Index, ISI | Pre, 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  The ISI will be used to assess self-reported levels of insomnia severity. Range is 0-28. Higher values represent higher levels of insomnia symptom severity.
Sleep diaries | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  Sleep diaries will be used to get daily information about: Sleep duration, sleep onset latency, wake after sleep onset, number of awakenings, bed time, rise time, time for final awakening before rise time, medication used, alchohol/drug use, variability. Individuals keep a record for at least 10 of 14 consecutive days.
Hospital Anxiety and Depression Scale, HADS | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  The HADS will be used to assess levels of anxiety and depression. The HADS comprises 14 items (higher values indicate higher symptom severity) pertaining to non-vegetative symptoms of anxiety and depression, which makes it a suitable measure of general psychological distress in populations likely to have physical comorbidities (e.g. general practice and liaison psychiatry settings).
Short Form-12, SF-12 | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  The SF-12 is an abbreviated version of the MOS 36-item short-form health survey (SF-36), and measures the individuals' perceived physical and mental health status. The SF-12 is scored using the recommended MOS software program that creates two summary scores, mental health (MCS12), and physical health (PCS12). The scores are represented as T-scores that are linear transformations with a mean of 50 and a standard deviation of 10 in the general U.S. population.
Dysfunctional Beliefs About Sleep scale, DBAS | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  The DBAS is a self-report questionnaire designed to identify maladaptive sleep- and insomnia-related cognitions. Patients are given a list of 16 statements reflecting different beliefs and attitudes about sleep, and they are asked to indicate on a 10-point scale how much they agree with the statements. Higher scores indicate higher levels of endorsement of beliefs.
Chalder Fatigue Questionnaire, CFQ | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  The CFQ comprises 11 items addressing physical and psychological fatigue, and two items addressing the duration and the intensity of fatigue complaints. Higher values indicate higher levels of fatigue.
The Bergen Insomnia Scale, BIS | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  The BIS comprises six items that assesses symptoms of insomnia based on the insomnia criteria found in the Diagnostic and Statistical Manual of Mental Disorders-IV-TR (American Psychiatric Association). Higher values indicate higher levels of insomnia severity.
Brief Horne-Östberg Morningness-Eveningness Questionnaire, MEQ | Pre, 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  The MEQ is the most widely used measure of chronotype (so-called 'morningness' or 'eveningness'), and gives an indication of the respondents preferred (as opposed to actual) rise-time and bed-time. Higher scores indicate higher levels of morningness.
Physical health | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  A 20-item checklist of common medical conditions and any impact on work or personal life. Also used in the Helseundersøkelsen Nordtrøndelag study (the HUNT study).
Mental health | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  Presence of psychiatric conditions will be assessed with an 8-item checklist of common psychiatric conditions based on a template used for physical health in the Helseundersøkelsen Nordtrøndelag study (the HUNT study).
Pain site | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  A self-report checklist (yes/no) of nine sites on the body where one can experience pain.
Alcohol use disorders identification test - consumption , AUDIT-C | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  The AUDIT-C scale comprises of three items and will be used to assess the frequency and quantity of alcohol consumption where higher scores indicate higher levels of use.
Body Mass Index | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  Height will be recorded at baseline and weight will be recorded at baseline, post-intervention, 6 and 24 months to allow estimation of body mass index (kg/m^2) at these time points.
Physical activity | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  Level of self-reported physical activity is measured using six items (from the HUNT study) that assess frequency, intensity and duration of the activity.
National Insurance Administration (NIA) | Pre intervention, 12 months and 9 weeks after randomization, and 24 months and 9 weeks after randomization
  Objective data on days with sick leave will be determined with data from the NIA, a national Norwegian registry which records all periods of sick leave >13 days, as well as information on all disability pension awards.
Norwegian Patient Registry (NPR) | Pre intervention, 12 months and 9 weeks after randomization, and 24 months and 9 weeks after randomization
  Objective data on the use and type of specialist health care services will be determined using the NPR, a national Norwegian registry which contains information about all patients who are waiting for, or have received treatment, as outpatients in the specialist health service. The data retrieved from the NPR include diagnoses (according to ICD-10 criteria), name of health care provider, service use (e.g. outpatient appointments) and hospital admission and discharge dates.
Norwegian Prescription Database (NorPD) | Pre intervention, 12 months and 9 weeks after randomization, and 24 months and 9 weeks after randomization
  Medication use will be determined from NorPD, a national health register comprising information on all prescriptions dispensed at Norwegian pharmacies (since January 2004). The NorPD provides detailed information that will allow us to identify the medication, its class, and information on dispensed prescriptions (which can be used as a proxy for medication consumption).
Help seeking behavior | 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  A self-report 10-item questionnaire that records what help or treatments that have been sought.
Medication use | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  Free text where participants report reason for medication use, dosage, timing, and adherence.
Use of health care services | Pre, 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  Subjective reports of health care service use will be assessed with 5 items recording use of primary and secondary health services.
Absence from work and loss of productivity | Pre, 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  A self-report 7 item questionnaire that assess absence from work and loss of productivity due to health problems.
Impact of health problems on productivity | Pre, 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  2 items recording self-perceptions of any negative effects of health status on work or leisure activities.
Internet intervention evaluation | 9 weeks after randomization (post assessment), and 24 months follow-up (24 months and 9 weeks after randomization)
  The acceptability of online interventions after completion of the programs will be assessed with the Internet intervention evaluation which comprises two questionnaires used in SHUTi research: the Internet Intervention Utility Questionnaire (UQ) and the Internet Intervention Impact Questionnaire (IQ).
Electronic Media Use | Pre, 9 weeks after randomization (post assessment), 6 months follow-up (6 months and 9 weeks after randomization), 24 months follow-up (24 months and 9 weeks after randomization)
  Self-report ratings of how much daily time participants spend, and how much time they spend while in bed, on different five different types of electronic media.
Negative Effects Questionnaire, NEQ | 24 months follow-up (24 months and 9 weeks after randomization)
  To assess views regarding the interventions, we will ask participants to complete the NEQ. The NEQ is a self-report measure that contains 32 items that are scored on a five point Likert-scale (0-4) where higher scores indicate higher levels of negative effects. After each item, the individual is asked whether they consider the effect to be caused by the treatment received or caused by other circumstances (yes/no), as well as one open-ended question.
Use of sleep strategies questionnaire | 24 months follow-up (24 months and 9 weeks after randomization)
  A self-report questionnaire has been developed in order to assess patients continued use of sleep strategies after the intervention. The questionnaire comprises 6 items assessing how many times each week the last month patients have used 6 different therapeutic techniques used in Cognitive Behavior Therapy for Insomnia (incl. kept a stable rise time, refrained from sleeping during daytime, used the bed and the bedroom only for sleeping, practiced sleep restriction, got out of the bed when unable to fall asleep within 15-20 minutes, and kept a sleep diary), how useful each technique was on a 0 to 10 scale where higher score indicates higher level of usefulness, and whether the patients have used the technique regularly since terminating treatment (yes/no).

OTHER OUTCOMES:
Salivary sample | Single sample 24 months and 9 weeks after randomization (depending on funding/ethics approval for this component of the study)
  Sample to be used to assess genetic factors (eg SNPs) as a putative moderator.

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Norwegian Institute of Public Health, Bergen
  - NTNU, Trondheim

REFERENCES:
- [Derived] Skoglund H, Sivertsen B, Kallestad H, Vedaa O. Digital cognitive behavioral therapy for insomnia for people with comorbid psychological distress: A large scale randomized controlled trial. Sleep Med. 2024 Sep;121:241-250. doi: 10.1016/j.sleep.2024.06.026. Epub 2024 Jun 28. PMID 39024778
- [Derived] Vestergaard CL, Vedaa O, Simpson MR, Faaland P, Vethe D, Kjorstad K, Langsrud K, Ritterband LM, Sivertsen B, Stiles TC, Scott J, Kallestad H. The effect of sleep-wake intraindividual variability in digital cognitive behavioral therapy for insomnia: a mediation analysis of a large-scale RCT. Sleep. 2021 Oct 11;44(10):zsab118. doi: 10.1093/sleep/zsab118. PMID 33964166
- [Derived] Vedaa O, Kallestad H, Scott J, Smith ORF, Pallesen S, Morken G, Langsrud K, Gehrman P, Thorndike FP, Ritterband LM, Harvey AG, Stiles T, Sivertsen B. Effects of digital cognitive behavioural therapy for insomnia on insomnia severity: a large-scale randomised controlled trial. Lancet Digit Health. 2020 Aug;2(8):e397-e406. doi: 10.1016/S2589-7500(20)30135-7. PMID 33328044
- [Derived] Kallestad H, Vedaa O, Scott J, Morken G, Pallesen S, Harvey AG, Gehrman P, Thorndike F, Ritterband L, Stiles TC, Sivertsen B. Overcoming insomnia: protocol for a large-scale randomised controlled trial of online cognitive behaviour therapy for insomnia compared with online patient education about sleep. BMJ Open. 2018 Aug 30;8(8):e025152. doi: 10.1136/bmjopen-2018-025152. PMID 30166311